CLINICAL TRIAL: NCT00853684
Title: Phase II Study of Oxaliplatin, Capecitabine and Endostar as First Line Treatment for Patients With Advanced Colorectal Cancer
Brief Title: Oxaliplatin, Capecitabine and Endostar as First Line Treatment for Patients With Advanced Colorectal Cancer
Acronym: OXCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200902024
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Advanced Colorectal Cancer
Keywords: Advanced Colorectal Cancer; Oxaliplatin; Capecitabine; Endostar; efficacy
MeSH Terms: interventions — Capecitabine; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oxaliplatin, capecitabine plus endostar (Experimental)
  Interventions: Drug: OXCE; Drug: Endostar

INTERVENTIONS:
Drug: OXCE — Oxaliplatin 130 mg/m2 iv drip D1, Capecitabine 1000 mg/m2 bid d1-14. Every three weeks.
  Other Names: Capecitabine(Xeloda®)
Drug: Endostar — Endostar 7.5 mg/m2 iv drip D1-14. Every 3 weeks.
  Other Names: Endostar (a recombinant human endostatin)

SUMMARY:
It is hypothesized that other anti-angiogenic agents such as endostar, may augment the effect of chemotherapy regimens in CRC. Endostar, a recombinant human endostatin which expressed and purified in E. coli, was approved by the SFDA for the treatment of non-small-cell lung cancer in 2005. Ling et al. found that endostar suppressed the VEGF-stimulated proliferation, migration, and tube formation of human umbilical vein endothelial cells (HUVECs) in vitro, and the antiangiogenic effects of endostar were correlated with the VEGF-triggered signaling. (Ling et al, 2007) A Chinese phase III clinical trial in advanced non-small-cell lung cancer, endostar--a new angiogenesis inhibitor prolonged the overall survival, time to progression and improved response rate. (Wang et al, 2005) Based on these results, the investigators design this phase II clinical trial of oxaliplatin, capecitabine and endostar as first line treatment, to evaluate whether endostar can bring survival benefits to patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
Among the different combination regimens of new drugs in CRC treatment, the combination of capecitabine and oxaliplatin seems especially attractive. Both drugs have a different and relatively mild toxicity profile. In phase II studies that used the recommended dose of XELOX (capecitabine 1000 mg/m2 twice daily on days 1-14 with intravenous oxaliplatin 130 mg/m2 on day 1 every 3 weeks), RRs were between 42% and 55%, with PFS times of 6.0 to 7.7 months, which showed that the XELOX combination was effective in the first-line treatment of patients with metastatic CRC. (Cassidy et al, 2004; Scheithauer et al, 2003)

Colorectal carcinomas (CRC) are characterised by enhanced VEGF expression and the corresponding high microvascular densities, indicating increased angiogenic activity and leading to worse patient survival.(Zheng et al, 2003; Des Guetz et al, 2006) Recently, the final results of XELOX-1/NO16966, a study of first line therapy, confirmed that bevacizumab+chemotherapy (XELOX or FOLFOX) was superior to chemotherapy alone in terms of PFS (HR 0.83; p=0.0023) although the OS data did not reach statistical significance (HR 0.89; p=0.0769). (Saltz et al, 2008)

The bevacizumab data provide a treatment option for patients with metastatic CRC based on VEGF inhibition. It is hypothesized that other anti-angiogenic agents such as endostar, may augment the effect of chemotherapy regimens in CRC. Endostar, a recombinant human endostatin which expressed and purified in E. coli, was approved by the SFDA for the treatment of non-small-cell lung cancer in 2005. Ling et al. found that endostar suppressed the VEGF-stimulated proliferation, migration, and tube formation of human umbilical vein endothelial cells (HUVECs) in vitro, and the antiangiogenic effects of endostar were correlated with the VEGF-triggered signaling. (Ling et al, 2007) A Chinese phase III clinical trial in advanced non-small-cell lung cancer, endostar--a new angiogenesis inhibitor prolonged the overall survival, time to progression and improved response rate. (Wang et al, 2005) Based on these results, we design this phase II clinical trial of oxaliplatin, capecitabine and endostar as first line treatment, to evaluate whether endostar can bring survival benefits to patients with advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or recurrent colorectal tumors with no previous treatment for advanced disease.
* Age greater than or equal to 18 years.
* SWOG performance status 0-1.
* At least one measurable lesion according to the RECIST criteria which has not been irradiated (i.e. newly arising lesions in previously irradiated areas are accepted). Minimum indicator lesion size: > 10 mm measured by spiral CT or >20mm measured by conventional techniques.
* Have a negative serum pregnancy test within 7 days prior to initiation of chemotherapy (female patients of childbearing potential).
* Availability of tumor biopsy (paraffin embedded or fresh frozen) at the time of diagnosis and/or prior to study entry is required.
* Patients must agree to have a 20 cc blood sample drawn in addition to routine labs with each cycle of chemotherapy.

Exclusion Criteria:

* Pregnant or lactating woman.
* Life expectancy < 3 months.
* Serious, uncontrolled, concurrent infection(s) or illness(es)
* Any prior oxaliplatin treatment, with the exception of adjuvant therapy given > 12 months prior to the beginning of study therapy
* Prior unanticipated severe reaction to fluoropyrimidine therapy, known hypersensitivity to 5-fluorouracil, or known DPD deficiency
* Prior unanticipated severe reaction or hypersensitivity to platinum based compounds.
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Current, recent (within 4 weeks of first infusion on this study) or planned participation in an investigational drug study.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) within the last 6 months.
* History of clinically significant interstitial lung disease and/or pulmonary fibrosis.
* History of persistent neurosensory disorder including but not limited to peripheral neuropathy.
* Presence of central nervous system or brain mets.
* Major surgery, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Any of the following laboratory values:

  * Abnormal hematologic values (neutrophils < 1.5 x 109/L, platelet count < 100 x 109/L)
  * Urine protein: creatinine ratio >/= 1.0 Impaired renal function with estimated creatinine clearance < 30 ml/min as calculated with Cockroft et Gault equation:
  * Serum bilirubin > 1.5 x upper normal limit. ALT, AST > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases)
  * Alkaline phosphatase > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases or > 10 x upper normal limit in the case of bone disease)
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Blood pressure > 150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* History of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 28 days prior to Day 0.
* Serious, non-healing wound, ulcer or bone fracture
* Carcinoma of any histology in close proximity to a major vessel, cavitation or history of hemoptysis.
* Completion of previous adjuvant chemotherapy regimen < four weeks prior to the start of study treatment (within six weeks of study treatment for mitomycin C and nitroureas), or with related toxicities unresolved prior to the start of study treatment.
* Karnofsky performance status <60.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 6 months

SECONDARY OUTCOMES:
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Cao, MD, Study Chair — Department of Oncology, Ruijin Hospital, Medical School of Shanghai Jiaotong University
Locations (1):
- Department of Oncology, Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Sun L, Ye HY, Zhang YH, Guan YS, Wu H. Epidermal growth factor receptor antibody plus recombinant human endostatin in treatment of hepatic metastases after remnant gastric cancer resection. World J Gastroenterol. 2007 Dec 7;13(45):6115-8. doi: 10.3748/wjg.v13.45.6115. PMID 18023113
- [Background] Xu F, Ma Q, Sha H. Optimizing drug delivery for enhancing therapeutic efficacy of recombinant human endostatin in cancer treatment. Crit Rev Ther Drug Carrier Syst. 2007;24(5):445-92. doi: 10.1615/critrevtherdrugcarriersyst.v24.i5.20. PMID 18197781